CLINICAL TRIAL: NCT01960257
Title: A Pilot Clinical Trial Characterizing Use of Ingestion Sensor Enabled Rifamate in Comparison to Directly Observed Therapy for the Treatment of Tuberculosis
Brief Title: Wirelessly Observed Therapy in Comparison to Directly Observed Therapy for the Treatment of Tuberculosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Proteus Digital Health, Inc. (Industry)
Responsible Party: Principal Investigator, Sara H. Browne, MD, MPH, Staff Research Associate, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AHF TB 001
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Tuberculosis
Keywords: tuberculosis; tuberculosis treatment; wirelessly observed therapy; proteus digital health; digital health feedback system
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHFS with IS-RM (Experimental): Digital Health Feedback System (DHFS) Rifamate (combination of isoniazid 150 mg and rifampin 300 mg) over-encapsulated with ingestion sensor - 2 capsules orally daily (QD) administered orally preferably on an empty stomach first thing in the morning for 10-16 weeks, depending on time left to complete TB treatment.
  Interventions: Device: Digital Health Feedback System
- SOC DOT (Active Comparator): Isoniazid 300 mg -1 tablet orally QD plus rifampin 300 mg - 2 capsules orally QD, OR Rifamate (combination of isoniazid 150 mg and rifampin 300 mg) - 2 capsules orally QD preferably on an empty stomach first thing in the morning for 10-16 weeks, depending on time left to complete TB treatment.
  Interventions: Other: SOC DOT

INTERVENTIONS:
Device: Digital Health Feedback System — This intervention uses an ingestion sensor and a wearable sensor (worn as a patch on the skin), which are new technologies approved by the FDA, to collect information about patients taking their TB medications. The wearable sensor records information, which is uploaded wirelessly to a mobile device and then to a secure computer. Together the sensors and the mobile device transmitting the information to the study computer are called a digital health feedback system (DHFS), which provides information about when patients have taken their TB medications.
  Other Names: DHFS
  Arms: DHFS with IS-RM
Other: SOC DOT
  Arms: SOC DOT

SUMMARY:
This study uses an ingestion sensor and a wearable sensor (worn as a patch on the skin), which are new Proteus Digital Health (PDH) technologies approved by the FDA, to collect information about patients taking their TB medications. The wearable sensor records information, which is uploaded wirelessly to a mobile device and then to a secure computer. Together the sensors and the mobile device transmitting the information to the study computer are called a digital health feedback system (DHFS), which gives healthcare providers information about when patients have taken their TB medications. The advantage of the DHFS is that patients can take their medication where and when it is convenient for them, and do not have to wait for a nurse to directly observe them taking their medication.

The purpose of this study is to find out if using these new technologies works as well as the standard method of observing in person when patients take their TB medications. This study will also look at the costs of using a DHFS for TB medications, what patients and healthcare providers think about using it, and other factors that can determine when one approach works better than another.

This study has two parts. For the first part of the study (Step I), patients will have an initial screening visit and then, in one two-week period, they will have 4 study visits at the UCSD AntiViral Research Center (AVRC) and routine visits from Public Health Services (PHS) workers. This part of the study is designed to confirm that the DHFS is working correctly and is accurately collecting information about each dose of medication that patients take, and to understand what patients and healthcare providers think about using the DHFS.

If patients are eligible for the second part of the study (Step II) and want to continue, that will last another 8-14 weeks with an additional 4 study visits at the AVRC. In the second part of the study, patients will be randomized into one of the following two groups.

Group 1: TB treatment is monitored by continued use of the DHFS

Group 2: TB treatment is monitored by the standard methods used by PHS (DOT)

The second part of the study is designed to compare these two methods of observing patients taking their TB medications, what the relative costs of these methods are , and the perception by patients and/or healthcare providers of the ease of use of the novel technology.

DETAILED DESCRIPTION:
PHARMACOKINETIC (PK) SUBSTUDY

The purpose of the PK substudy is to prospectively evaluate the pharmacokinetic parameters of isoniazid (INH) and rifampin (RIF) concentrations derived from dosing with Rifamate when given in native format compared to over encapsulated, ingestion sensor-enabled format.

The UCSD substudy aims to co-enroll 12 patients with Phase 1- the two-week investigation period of the characteristics of use of DHFS and patient acceptability. These subjects will be randomized to start on either Phase 1 or on two weeks of native Rifamate followed by 24-hour PK sampling.

ELIGIBILITY:
Inclusion Criteria

* Basic competency in understanding written and verbal information as it applies to DHFS use.
* Persons undergoing treatment for TB that includes at least isoniazid and rifampin at the time of entry to Phase 1; of note, patients must be sputum smear negative at the time of study entry.
* Laboratory values obtained by screening laboratories within 30 days of entry:

  * Absolute neutrophil count (ANC) >= 1,000/mm3.
  * Hemoglobin >= 9.0 g/dL.
  * Platelet count >= 75,000/mm3.
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase <= 3 x ULN.
  * Total bilirubin <= 1.5 x ULN and direct bilirubin.
* Females of childbearing potential must agree to use contraception throughout the study period.
* Men and women age >= 18 years.
* Eligible for anti-mycobacterial medications and in possession of prescriptions for isoniazid and rifampin, or Rifamate, as appropriate.
* Willing to follow all protocol requirements.
* Ability to use mobile device per investigator determination, and to wear PDH wearable sensor (i.e., no skin conditions precluding use).
* Ability and willingness of subjects to give written informed consent.

Exclusion Criteria

* Female who is pregnant or breast-feeding, or of childbearing potential and has a tuberculin positive test at screening and disagrees to use contraception throughout the study period.
* Use of any of the prohibited medications or other non-informed medications within 30 days of study entry.
* Known hypersensitivity to any of the study drugs.
* Known sensitivity to skin adhesives.
* Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 30 days prior to study entry (Day 0).
* Evidence of any anti-mycobacterial resistance, clinical or genetic, prior to study entry. Resistance testing results must be available for review by the site investigator and study protocol team prior to enrollment to ensure that no exclusionary resistance exists.
* Active drug or alcohol use, or dependence, or other conditions that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-10-25 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Browne, MD, MPH, Study Chair — University of California, San Diego
Locations (2):
- United States (2):
  - UCSD AntiViral Research Center, San Diego, California
  - San Diego County Public Health Services, San Diego, California

REFERENCES:
- [Derived] Browne SH, Umlauf A, Tucker AJ, Low J, Moser K, Gonzalez Garcia J, Peloquin CA, Blaschke T, Vaida F, Benson CA. Wirelessly observed therapy compared to directly observed therapy to confirm and support tuberculosis treatment adherence: A randomized controlled trial. PLoS Med. 2019 Oct 4;16(10):e1002891. doi: 10.1371/journal.pmed.1002891. eCollection 2019 Oct. PMID 31584944

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Stage 1, 92 participants screened, 77 were enrolled in WOT+ SOC DOT. Excluded from stage 2, n=16: 12 only participated in PK substudy, 3 withdrew consent and 1 withdrew due to AE.
  Stage 2, 61 participants enrolled and were divided into 2 arms, 41 in WOT, and 20 in DOT.
Groups:
- WOT+ SOC DOT: Digital Health Feedback System (DHFS) Rifamate (combination of isoniazid 150 mg and rifampin 300 mg) co-encapsulated with ingestion sensor - 2 capsules orally daily (QD) administered orally preferably on an empty stomach first thing in the morning for 10-16 weeks, depending on time left to complete TB treatment.
  Digital Health Feedback System: This intervention uses an ingestion sensor and a wearable sensor (worn as a patch on the skin), which are new technologies approved by the FDA, to collect information about patients taking their TB medications. The wearable sensor records information, which is uploaded wirelessly to a mobile device and then to a secure computer. Together the sensors and the mobile device transmitting the information to the study computer are called a digital health feedback system (DHFS), which provides information about when patients have taken their TB medications.
- Wirelessly Observed Therapy (WOT): IS-Rifamate (combination of isoniazid 150 mg and rifampin 300 mg) co-encapsulated with ingestion sensor - 2 capsules orally daily (QD) administered orally preferably on an empty stomach first thing in the morning for 10-16 weeks, depending on time left to complete TB treatment.
- Directly Observed Therapy (DOT): Isoniazid 300 mg -1 tablet orally QD plus rifampin 300 mg - 2 capsules orally QD, OR Rifamate (combination of isoniazid 150 mg and rifampin 300 mg) - 2 capsules orally QD preferably on an empty stomach first thing in the morning for 10-16 weeks, depending on time left to complete TB treatment.
  SOC DOT
Period: Stage 1 (1-3 Weeks)
Arm/Group | WOT+ SOC DOT | Wirelessly Observed Therapy (WOT) | Directly Observed Therapy (DOT)
Started | 77 | 0 | 0
Completed | 61 | 0 | 0
Not Completed | 16 | 0 | 0
Not completed — Only participated in PK Substudy | 12 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Stage 2(1-4 Months, Not to Exceed 12wks)
Arm/Group | WOT+ SOC DOT | Wirelessly Observed Therapy (WOT) | Directly Observed Therapy (DOT)
Started | 0 | 41 | 20
Completed | 0 | 41 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ALL PARTICIPANTS: Digital Health Feedback System (DHFS) Rifamate (combination of isoniazid 150 mg and rifampin 300 mg) co-encapsulated with ingestion sensor - 2 capsules orally daily (QD) administered orally preferably on an empty stomach first thing in the morning for 10-16 weeks, depending on time left to complete TB treatment.
  Isoniazid 300 mg -1 tablet orally QD plus rifampin 300 mg - 2 capsules orally QD, OR Rifamate (combination of isoniazid 150 mg and rifampin 300 mg) - 2 capsules orally QD preferably on an empty stomach first thing in the morning for 10-16 weeks, depending on time left to complete TB treatment.
  SOC DOT
  Digital Health Feedback System: This intervention uses an ingestion sensor and a wearable sensor (worn as a patch on the skin), which are new technologies approved by the FDA, to collect information about patients taking their TB medications. The wearable sensor records information, which is uploaded wirelessly to a mobile device and then to a secure computer. Together the sensors and the mobile device transmitting the information to the study computer are called a digital health feedback system (DHFS), which provides information about when patients have taken their TB medications.
Arm/Group | ALL PARTICIPANTS
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Each row represents data collected for a particular group based on treatment assignment.
  years
    Stage 1 | 43 (17)
    Stage 2 WOT: number analyzed (Participants) | 41
    Stage 2 WOT | 41 (16)
    Stage 2 DOT: number analyzed (Participants) | 20
    Stage 2 DOT | 45 (17)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Each row represents data collected for a particular group based on treatment assignment.
  Participants
    Stage 1: Female | 33
    Stage 1: Male | 44
    Stage 2 WOT: number analyzed (Participants) | 41
    Stage 2 WOT: Female | 20
    Stage 2 WOT: Male | 21
    Stage 2 DOT: number analyzed (Participants) | 20
    Stage 2 DOT: Female | 8
    Stage 2 DOT: Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Each row represents data collected for a particular group based on treatment assignment.
  Participants
    Stage 1: Hispanic or Latino | 38
    Stage 1: Not Hispanic or Latino | 36
    Stage 1: Unknown or Not Reported | 3
    Stage 2 WOT: number analyzed (Participants) | 41
    Stage 2 WOT: Hispanic or Latino | 21
    Stage 2 WOT: Not Hispanic or Latino | 18
    Stage 2 WOT: Unknown or Not Reported | 2
    Stage 2 DOT: number analyzed (Participants) | 20
    Stage 2 DOT: Hispanic or Latino | 11
    Stage 2 DOT: Not Hispanic or Latino | 8
    Stage 2 DOT: Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Each row represents data collected for a particular group based on treatment assignment.
  Participants
    Stage 1: American Indian or Alaska Native | 0
    Stage 1: Asian | 32
    Stage 1: Native Hawaiian or Other Pacific Islander | 1
    Stage 1: Black or African American | 1
    Stage 1: White | 30
    Stage 1: More than one race | 0
    Stage 1: Unknown or Not Reported | 13
    Stage 2 WOT: number analyzed (Participants) | 41
    Stage 2 WOT: American Indian or Alaska Native | 0
    Stage 2 WOT: Asian | 17
    Stage 2 WOT: Native Hawaiian or Other Pacific Islander | 1
    Stage 2 WOT: Black or African American | 0
    Stage 2 WOT: White | 14
    Stage 2 WOT: More than one race | 0
    Stage 2 WOT: Unknown or Not Reported | 9
    Stage 2 DOT: number analyzed (Participants) | 20
    Stage 2 DOT: American Indian or Alaska Native | 0
    Stage 2 DOT: Asian | 8
    Stage 2 DOT: Native Hawaiian or Other Pacific Islander | 0
    Stage 2 DOT: Black or African American | 0
    Stage 2 DOT: White | 8
    Stage 2 DOT: More than one race | 0
    Stage 2 DOT: Unknown or Not Reported | 4
Employment status: full-time/part time [Count of Participants; unit: Participants] — Population: Each row represents data collected for a particular group based on treatment assignment.
  Participants
    Stage 1: Full-time | 21
    Stage 1: Part-time | 8
    Stage 1: Unemployed | 32
    Stage 1: Retired | 4
    Stage 1: Unable to work (disabled) | 12
    Stage 2 WOT: number analyzed (Participants) | 41
    Stage 2 WOT: Full-time | 12
    Stage 2 WOT: Part-time | 5
    Stage 2 WOT: Unemployed | 18
    Stage 2 WOT: Retired | 0
    Stage 2 WOT: Unable to work (disabled) | 6
    Stage 2 DOT: number analyzed (Participants) | 20
    Stage 2 DOT: Full-time | 6
    Stage 2 DOT: Part-time | 2
    Stage 2 DOT: Unemployed | 7
    Stage 2 DOT: Retired | 1
    Stage 2 DOT: Unable to work (disabled) | 4

OUTCOME MEASURES:

1. Primary Outcome: Step 1: Positive Detection Accuracy (PDA)
Description: Determine positive detection accuracy (PDA, direct confirmation of TB medication ingestion) of the DHFS when compared to a healthcare worker witnessing actual TB medication ingestion.
Time Frame: 2 weeks
Population: Positive Detection Accuracy (PDA): PDA is defined as DHFS detection of the ingestion of a dose of IS-RM when compared to a witnessed ingestion of the same dose of medication.
Measure: Number (95% Confidence Interval); unit: percentage of DHFS detected doses
Groups:
- DHFS With IS-RM Plus SOC DOT: Initially all participants (n=77) received DHFS IS-RM in conjunction with witnessed medication doses (DOT) for 2-3 weeks to allow calculation of DHFS IS-RM PDA, and the 95% confidence interval (CI) was estimated using the bootstrap method with 10,000 samples.
Arm/Group | DHFS With IS-RM Plus SOC DOT
Number analyzed (Participants) | 77
percentage of DHFS detected doses | 99.3 [98.1 to 100]

2. Primary Outcome: Step 2: Percentage of Witnessed Doses
Description: Determine the percentage of witnessed doses by DHFS and standard of care (SOC), respectively.
Time Frame: 16 weeks
Population: Observation days
Measure: Number (95% Confidence Interval); unit: percentage of witnessed doses
Units Other Than Participants: Days
Groups:
- Wirelessly Observed Therapy (WOT): IS-Rifamate (combination of isoniazid 150 mg and rifampin 300 mg) co-encapsulated with ingestion sensor - 2 capsules orally daily (QD) administered orally preferably on an empty stomach first thing in the morning for 10-16 weeks, depending on time left to complete TB treatment.
  Digital Health Feedback System: This intervention uses an ingestion sensor and a wearable sensor (worn as a patch on the skin), which are new technologies approved by the FDA, to collect information about patients taking their TB medications. The wearable sensor records information, which is uploaded wirelessly to a mobile device and then to a secure computer. Together the sensors and the mobile device transmitting the information to the study computer are called a digital health feedback system (DHFS), which provides information about when patients have taken their TB medications.
- SOC DOT: Isoniazid 300 mg -1 tablet orally QD plus rifampin 300 mg - 2 capsules orally QD, OR Rifamate (combination of isoniazid 150 mg and rifampin 300 mg) - 2 capsules orally QD preferably on an empty stomach first thing in the morning for 10-16 weeks, depending on time left to complete TB treatment.
  SOC DOT
Arm/Group | Wirelessly Observed Therapy (WOT) | SOC DOT
Number analyzed (Participants) | 41 | 20
Number analyzed (Days) | 93 | 101
percentage of witnessed doses | 92.9 [89 to 96] | 63.1 [58 to 67]

3. Secondary Outcome: Characterize Subject Responses to Post-study Questionnaires to Collect Information Regarding Their Experience With the DHFS Using Summary Statistics.
Description: Subject responses regarding satisfaction with the DHFS were reported on post study questionnaires regarding their experience with the DHFS and the usability of the system, using summary statistics. Areas evaluated may include ease of use, time needed to use the system, negative impressions, and changes to quality of life. Analyses of individual questions as well as summary metrics across questions were explored.
  Percentage of participants who reported being comfortable replacing the patch on their own
Time Frame: 2-3 weeks
Population: Ease of use of the DHFS
Measure: Number; unit: percentage of participants
Groups:
- Stage 1: DHFS With IS-RM Plus SOC DOT: Initially all participants (n=77) received DHFS IS-RM in conjunction with witnessed medication doses (DOT) for 2-3 weeks to allow calculation of DHFS IS-RM PDA, and the 95% confidence interval (CI) was estimated using the bootstrap method with 10,000 samples.
- Stage 2: DHFS With IS-RM: n=41 participants were randomized to the Intervention Group that used DHFS with IS-RM without concurrent DOT for TB treatment monitoring
Arm/Group | Stage 1: DHFS With IS-RM Plus SOC DOT | Stage 2: DHFS With IS-RM
Number analyzed (Participants) | 71 | 41
percentage of participants | 75.3 | 92.8

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for 2 weeks in Stage 1 and up to 12 months in Stage 2, Through study completion, an average of 12 months, or similar.
Groups:
- WOT+ SOC DOT: Digital Health Feedback System (DHFS) Rifamate (combination of isoniazid 150 mg and rifampin 300 mg) over-encapsulated with ingestion sensor - 2 capsules orally daily (QD) administered orally preferably on an empty stomach first thing in the morning for 10-16 weeks, depending on time left to complete TB treatment.
  Digital Health Feedback System: This intervention uses an ingestion sensor and a wearable sensor (worn as a patch on the skin), which are new technologies approved by the FDA, to collect information about patients taking their TB medications. The wearable sensor records information, which is uploaded wirelessly to a mobile device and then to a secure computer. Together the sensors and the mobile device transmitting the information to the study computer are called a digital health feedback system (DHFS), which provides information about when patients have taken their TB medications.
- Wirelessly Observed Therapy (WOT): IS-enabled combination isoniazid 150 mg/rifampin 300 mg (IS-Rifamate) over-encapsulated with ingestion sensor - 2 capsules orally daily (QD) administered orally preferably on an empty stomach first thing in the morning for 10-16 weeks, depending on time left to complete TB treatment.
  Digital Health Feedback System: This intervention uses an ingestion sensor and a wearable sensor (worn as a patch on the skin), which are new technologies approved by the FDA, to collect information about patients taking their TB medications. The wearable sensor records information, which is uploaded wirelessly to a mobile device and then to a secure computer. Together the sensors and the mobile device transmitting the information to the study computer are called a digital health feedback system (DHFS), which provides information about when patients have taken their TB medications.
Arm/Group | WOT+ SOC DOT | Wirelessly Observed Therapy (WOT) | Directly Observed Therapy (DOT)
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/41 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/41 | 0/20
Other Adverse Events (participants affected / at risk) | 1/77 | 0/41 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WOT+ SOC DOT (N=77) | Wirelessly Observed Therapy (WOT) (N=41) | Directly Observed Therapy (DOT) (N=20)
Pruritus at patch site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT01960257/Prot_SAP_000.pdf